CLINICAL TRIAL: NCT04786535
Title: Crossover Study of Three Groups Comparing the Efficacy of Uremic Toxins Clearance of Expanded Hemodialysis With Two Hemodialysis Membranes for Conventional Hemodialysis and Hemodiafiltration
Brief Title: Efficacy of Uremic Toxins Clearance With Expanded Hemodialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: Baxter México (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: REF.2937
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: End Stage Renal Disease
Keywords: Uremic Toxins; Hemodiafiltration; Expanded Hemodialysis; High-Flux Conventional Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Hemodiafiltration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hemodiafiltration (Active Comparator)
  Interventions: Procedure: Hemodiafiltration
- Expanded hemodialysis (Experimental)
  Interventions: Procedure: Expanded Hemodialysis
- Conventional high-flux hemodialysis (Experimental)
  Interventions: Procedure: High-flux Conventional Hemodialysis

INTERVENTIONS:
Procedure: Expanded Hemodialysis — * Single-use Theranova 400 Dialyzer
  * Blood flow (Qb) minimum of 300 mL/min
  * Dialysis flow (Qd) 500 mL/min
  * Minimum therapy time of 4 hours
  * Ultrafiltration necessary to achieve dry weight
  Arms: Expanded hemodialysis
Procedure: High-flux Conventional Hemodialysis — * Single-use high-flux hemodialyzer
  * Blood flow (Qb) minimum of 300 mL/min
  * Dialysis flow (Qd) 500 mL/min
  * Minimum therapy time of 4 hours
  * Ultrafiltration necessary to achieve dry weight
  Arms: Conventional high-flux hemodialysis
Procedure: Hemodiafiltration — * Single-use high-flux hemodialyzer
  * Post-dilution mode
  * Minimum convective volume of 23 L
  * Blood flow (Qb) minimum of 300 mL/min
  * Dialysis flow (Qd) 700 mL/min
  * Minimum therapy time of 4 hours
  * Ultrafiltration necessary to achieve dry weight
  Arms: Hemodiafiltration

SUMMARY:
The aim of this study is to quantify the B2-microglobulin reduction rate based on the type of extracorporeal therapy (ET) used: HDx (expanded hemodialysis), HDc (high-flux conventional hemodialysis), or HDF (hemodiafiltration).

And to compare the magnitude of the B2-microglobulin reduction rate based on the type of extracorporeal therapy (ET) used: HDx, HDc, or HDF

DETAILED DESCRIPTION:
A controlled, randomized, crossover clinical trial is planned to compare the magnitude of the B2-microglobulin reduction rate in three different extracorporeal therapies (ETs): HDc, HDx, and HDF.

The selection of study participants will be consecutive and for convenience

This study will be divided into six periods: three treatment periods (one for each therapy to be compared) and three of "washout" periods (interspersed between the treatment periods). The treatment periods will last four weeks (12 ET sessions, three per week) and will be preceded by a one-week washout period (three ET sessions)

After inclusion in the protocol, participants will be randomly assigned (with the help of a table of random numbers) to one of three ETs to be evaluated (HDc, HDx, or HDF). Afterwards, the first washout period will begin with high-flow conventional hemodialysis (HDc). At the end of the first washout period, the ET randomly assigned to one of three ETs to be evaluated (HDc, HDx, or HDF), following the sequence: Washout 1 -> Period 1 (HDC, HDx, or HDF) -> Washout 2 -> Period 2, etc.

For each period of ET, there will be two sampling times: baseline and final

Blood samples will be obtained through the arterial port of the extracorporeal circuit, at the beginning and at the end of the ET session. The "slow flow" method will be used (UF: 0 mL/min, Qd: 0 mL/min, and Qb: 100 mL/min, for 30 seconds, before extracting the sample from the arterial port) (24). Blood samples will be collected in dry tubes (without anticoagulant) and centrifuged for 10 minutes at 3,000 RPM. The supernatant will be divided into three aliquots and stored at -70°C for further processing.

To calculate sample size, the formula for a noninferiority study was used (Pharmaceutical statistics. 2016;15(1):80-9), which is detailed below:

n= ((r+1) (Z_(1-β)+Z_(1-α) )^2 σ^2)/(r((μ_A-μ_B )-d_NI )^2 )

The terms above, are substituted with values obtained from the publication of Kirsch et al. (Nephrol Dial Transplant. 2017 Jan 1;32(1):165-172) as follows:

Objective: Non-inferiority (Ho µA - µB ≤ -dNI vs. µA - µB > -dNI) Outcome: B2-microglobulin reduction rate. r: allocation ratio by group:1 beta: type II error (90% power):1.2816 alpha: type I error (level of significance 5%):1.960 (variance in the population):1.33 µA - µB (magnitude of the observed effect):80.6 - 78.5 = 2.1 dNI (non-inferiority limit): 3.5

n= ((1+1) (1.2816+1.960)^2 〖(1.33)〗^2)/(1((2.1)-3.5)^2 )= 19, the investigators estimate a 20 % loss in the follow-up , then investigators consider a sample size of n = 23 patients

The nominal variables will be presented in frequencies and proportions. Continuous numerical variables will be analyzed using the Kolmogorov-Smirnov "Z" test to determine their distribution. The results will be shown as the means ± standard deviation in case of normal distribution and as a median with minimum and maximum limits for variables with non-normal distribution.

The total serum concentration of the biochemical variables in general as well as the uremic toxins will be analyzed. Additionally, the reduction rate and purification of the uremic toxins will be analyzed.

The analyses of the inter- and intra-group differences will be performed using the one-way multiple comparisons (ANOVA) method. Post hoc analysis using the Bonferroni method will be used in cases where the groups present a normal distribution; otherwise, the Kruskal-Wallis method will be used. A result with a p < 0.05 will be considered significant

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Anuric patients (residual urinary volume ≤ 100 mL/24 h)
* Intermittent chronic hemodialysis (three sessions per week, of 3.5 to 4 hours each)
* Without modification of their prescription in the last three months
* Functional arteriovenous fistula, indwelling vascular access (Qb ≥ 300 mL/min), or both
* Letter of acceptance to enter the protocol and a signed informed consent.

Exclusion Criteria:

* Under 18 years
* Active intake or intake in the last six months of immunosuppressants or systemic steroids
* Active autoimmune disease
* Evidence of active systemic infectious event at the time of inclusion or two weeks prior
* Diagnosis of neoplasia or active oncological disease
* Hypoalbuminemia (< 3.2 g/dL)
* Pregnancy or lactation
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-09-06 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
B2-microglobulin reduction rate | At final of each period of ET (4 weeks)
  B2-microglobulin reduction rate based on the type of extracorporeal therapy (ET) used: HDx, HDc, or HDF.

SECONDARY OUTCOMES:
Urea reduction rate | At final of each period of ET (4 weeks)
  Urea reduction rate based on the type of extracorporeal therapy (ET) used: HDx, HDc, or HDF.
Phosphorus reduction rate | At final of each period of ET (4 weeks)
  Phosphorus reduction rate based on the type of extracorporeal therapy (ET) used: HDx, HDc, or HDF.
Interleukin 6 reduction rate | At final of each period of ET (4 weeks)
  Interleukin 6 reduction rate based on the type of extracorporeal therapy (ET) used: HDx, HDc, or HDF.
P-cresol reduction rate | At final of each period of ET (4 weeks)
  P-cresol reduction rate based on the type of extracorporeal therapy (ET) used: HDx, HDc, or HDF.
Tumor necrosis factor-a reduction rate | At final of each period of ET (4 weeks)
  Tumor necrosis factor-a reduction rate based on the type of extracorporeal therapy (ET) used: HDx, HDc, or HDF.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Correa-Rotter, MD, Principal Investigator — Head Departament of Nephrology and Mineral Metabolism,
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belmouaz M, Diolez J, Bauwens M, Duthe F, Ecotiere L, Desport E, Bridoux F. Comparison of hemodialysis with medium cut-off dialyzer and on-line hemodiafiltration on the removal of small and middle-sized molecules . Clin Nephrol. 2018 Jan;89 (2018)(1):50-56. doi: 10.5414/CN109133 . PMID 28853700
- [Background] Ronco C. The Rise of Expanded Hemodialysis. Blood Purif. 2017;44(2):I-VIII. doi: 10.1159/000476012. Epub 2017 May 10. PMID 28486230
- [Background] Ronco C, Marchionna N, Brendolan A, Neri M, Lorenzin A, Martinez Rueda AJ. Expanded haemodialysis: from operational mechanism to clinical results. Nephrol Dial Transplant. 2018 Oct 1;33(suppl_3):iii41-iii47. doi: 10.1093/ndt/gfy202. PMID 30281134
- [Background] Zickler D, Schindler R, Willy K, Martus P, Pawlak M, Storr M, Hulko M, Boehler T, Glomb MA, Liehr K, Henning C, Templin M, Trojanowicz B, Ulrich C, Werner K, Fiedler R, Girndt M. Medium Cut-Off (MCO) Membranes Reduce Inflammation in Chronic Dialysis Patients-A Randomized Controlled Clinical Trial. PLoS One. 2017 Jan 13;12(1):e0169024. doi: 10.1371/journal.pone.0169024. eCollection 2017. PMID 28085888
- [Background] Kirsch AH, Lyko R, Nilsson LG, Beck W, Amdahl M, Lechner P, Schneider A, Wanner C, Rosenkranz AR, Krieter DH. Performance of hemodialysis with novel medium cut-off dialyzers. Nephrol Dial Transplant. 2017 Jan 1;32(1):165-172. doi: 10.1093/ndt/gfw310. PMID 27587605